CLINICAL TRIAL: NCT01461395
Title: A Non-invasive Method to Assess DNA Damage in Individual Sperm
Brief Title: Polscope Sperm: A Non-invasive Method to Assess DNA Damage in Individual Sperm
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 107209
Record Dates: First submitted 2011-02-02; First posted 2011-10-28 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: DNA Damage; Other Complications Associated With Artificial Fertilization
Keywords: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sperm
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to find a non-invasive way to discover DNA (deoxyribonucleic acid, which is the genetic material inside your cells) alterations in the sperm's head, in the near future leading us to choose the "good sperm" in a simplified manner. This could then increase chances of a successful in-vitro fertilization (IVF) treatment when there are sperm abnormalities.

DETAILED DESCRIPTION:
If you take part in this study,

1. Your physician is asking you to provide a semen sample as you already would. The sample will be taken to the IVF lab which would occur if you were not involved in this research. The part that would be thrown away is then further analyzed under a polarized light microscope. The sample is exposed to ultraviolet (UV) light for a period of 20 minutes after which it is analyzed under the microscope again, looking for any changes when compared the sample that was not exposed to UV light. The sample is then discarded.
2. Your name will be removed from the sample after the regular semen analysis is done; therefore there will be no way of associating the research results with you. No information will be needed from you and you will not be contacted in the future regarding this research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* provide informed consent
* Already providing a semen sample as routine therapy in IVF

Exclusion Criteria:

-unable to provide informed consent

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IVF patients already undergoing therapy and providing a semen sample for sperm count
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celso Silva, M.D, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida South Tampa Center, Tampa, Florida, United States

REFERENCES:
- See also: USF Clinical Trials — http://www.research.usf.edu/cs/irb.htm